CLINICAL TRIAL: NCT00000236
Title: Buprenorphine Pharmacology Related to Addiction Treatment
Brief Title: Buprenorphine Pharmacology Related to Addiction Treatment - 18
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-18; R01-06969-18
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2002-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to examine the interactions between buprenorphine and naltrexone, and to assess how they may directly impact the clinical issues involving: transferring patients from buprenorphine to naltrexone, developing a non-abusable form of buprenorphine, and enhancing patient acceptability of naltrexone.

ELIGIBILITY:
Please contact site for information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0

PRIMARY OUTCOMES:
Drug use
Opioid agonist effects
Opiate withdrawal
Psychological changes in: pupil diameter, blood pressure, heart rate, respiration

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States